CLINICAL TRIAL: NCT00281658
Title: A Randomized, Multicenter, Double-Blind, Placebo-Controlled, Phase III Study of Lapatinib (GW572016) in Combination With Paclitaxel Versus Paclitaxel Plus Placebo in Subjects With ErbB2 Amplified Metastatic Breast Cancer
Brief Title: Study In Women And Men With Metastatic Breast Cancer That Have Overexpression Of ErbB2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EGF104535; CLAP016A2302 (Other: Novartis)
Record Dates: First submitted 2006-01-23; First posted 2006-01-25 (Estimated); Results first posted 2011-06-01 (Estimated); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Neoplasms, Breast
Keywords: ErbB2 positive; human epidermal growth factor receptor 2 positive (Her2+); metastatic breast cancer; Fluorescence in situ hybridization (FISH) positive; Stage IV
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Paclitaxel and Lapatinib (Blinded) (Experimental): Paclitaxel and Lapatinib (Blinded)
  Interventions: Drug: Lapatinib (GW572016) oral tablets; Drug: Paclitaxel infusion
- Paclitaxel and Placebo (Blinded) (Active Comparator): Paclitaxel and Placebo (Blinded)
  Interventions: Drug: Paclitaxel infusion; Drug: Placebo
- Open Label - Monotherapy (Extension Phase) (Other): Open Label - Monotherapy (Lapatinib)
  Interventions: Drug: Lapatinib (GW572016) oral tablets
- Open Label - Combination Therapy (Extension Phase) (Other): Open Label - Combination Therapy (Lapatinib and Paclitaxel)
  Interventions: Drug: Lapatinib (GW572016) oral tablets; Drug: Paclitaxel infusion

INTERVENTIONS:
Drug: Lapatinib (GW572016) oral tablets — 1500 mg oral daily continuously
  Arms: Open Label - Combination Therapy (Extension Phase); Open Label - Monotherapy (Extension Phase); Paclitaxel and Lapatinib (Blinded)
Drug: Paclitaxel infusion — Paclitaxel 80 mg/m2 every 3 weeks, 4th week rest for minimum 6 months
  Arms: Open Label - Combination Therapy (Extension Phase); Paclitaxel and Lapatinib (Blinded); Paclitaxel and Placebo (Blinded)
Drug: Placebo — Paclitaxel Matching Placebo
  Arms: Paclitaxel and Placebo (Blinded)

SUMMARY:
This was a randomized, double-blind, placebo-controlled, multicenter, Phase III study to evaluate and compare the efficacy and safety of Lapatinib + Paclitaxel versus Placebo + Paclitaxel in men and women with ErbB2 amplified metastatic (Stage IV) breast cancer who had not received prior therapy for metastatic disease.

DETAILED DESCRIPTION:
Subjects were randomized to receive either Lapatinib (1500 mg once daily) + Paclitaxel (80 mg/m2 IV weekly for 3 weeks every 4 weeks) or Placebo (once daily) + Paclitaxel (80 mg/m2 IV weekly for 3 weeks every 4 weeks).

Subjects who progressed while on study and were on the placebo+paclitaxel arm were permitted to enter an extension phase of open label monotherapy therapy with lapatinib or open label combination therapy with lapatinib+paclitaxel and followed for response, progression and survival.

Based on the positive results in the primary analysis, Protocol Amendment 02 (dated 09 May 2011) discontinued further entry into the lapatinib monotherapy extension phase, and ongoing subjects taking placebo were permitted to replace it with open label lapatinib therapy (with or without continued paclitaxel therapy).

Following the primary Overall Survival (OS) analysis and subsequent implementation of Protocol Amendment 03, subjects who were still receiving active treatment entered the Long-term follow-up (LTFU) phase of the study. Reporting requirements in the LTFU phase were limited to Adverse events of special interest (AESI), Serious adverse events (SAEs) and pregnancy, and the subjects continued to receive treatment until the occurrence of unacceptable toxicity or disease progression (as determined by the investigator) or permanent withdrawal from treatment for any reason. Subjects who were no longer receiving active treatment were withdrawn from the study.

ELIGIBILITY:
Inclusion criteria:

* Signed informed consent;
* Male or female ≥18 years;
* Histologically confirmed invasive breast cancer with stage IV disease; If the disease is restricted to a solitary lesion, its neoplastic nature should be confirmed by cytology or histology.
* Documented amplification of ErbB2 by fluorescence in situ hybridization (FISH) in primary or metastatic tumor tissue by the central laboratory for randomization into the study;
* If a taxane was administered in the neoadjuvant or adjuvant setting, progression must have occurred >12 months after completion of this treatment and the patient recovered from all associated toxicities;
* Measurable lesion(s) according to RECIST (Response Evaluation Criteria in Solid Tumors);
* Radiotherapy as palliative treatment for painful metastatic disease is permitted but must have been stopped within 2 weeks prior to initiation of any investigational treatment. All subjects must have recovered from all radiotherapy related toxicities prior to initiation of any investigational treatment. The site of radiotherapy must not be used as a site of measurable disease;
* Bisphosphonate therapy for bone metastases and is allowed; however, treatment must be initiated prior to the first dose of investigational treatment. Prophylactic use of bisphosphonates in subjects without bone disease is not permitted, except for the treatment of osteoporosis;
* For those patients whose disease is ER+ and/or PR+ the following criteria should be met:

Patients with visceral disease that requires chemotherapy (eg., patients with liver or lung metastases) Rapidly progressing or life threatening disease, as determined by the investigator Patients who received hormonal therapy and are no longer benefiting from this therapy and the hormonal treatment must have been stopped before the first dose of investigational treatment;

* Cardiac ejection fraction within institutional range of normal as measured by echocardiogram. MUGA scans will be accepted in cases where an echocardiogram cannot be performed or is inconclusive;
* ECOG Performance Status of 0 to 1;
* Life expectancy of ≥ 12 weeks;
* Able to swallow and retain oral medication;
* Archived tumor tissue available for testing;
* Women and men with potential to have children must be willing to practice acceptable methods of birth control during the study;
* Willing to complete all screening assessments as outlined in the protocol;
* Adequate organ function as defined in Table 1 Baseline Laboratory Values;

Exclusion Criteria:

* Pregnant or lactating females at anytime during the study
* Subjects with only non-measurable metastatic sites of disease per RECIST, (e.g. bone metastases, pleural effusion, or ascites, etc. (Refer to Section 5.3 Efficacy for list sites considered to be non-measurable disease.);
* Received prior chemotherapy, immunotherapy, biologic therapy, or anti-ErbB1/ErbB2 therapy for metastatic disease.
* Prior therapy with an ErbB1 and/or ErbB2 inhibitor, other than trastuzumab in the adjuvant setting. If trastuzumab was administered in the adjuvant setting, then > 12 months must have elapsed since completion of trastuzumab therapy;
* Planned concurrent anti-cancer therapy (chemotherapy, radiation therapy, immunotherapy, biologic therapy, hormonal therapy) while taking investigational treatment;
* Unresolved or unstable, serious toxicity from prior administration of another investigational drug and/or of prior cancer treatment;
* Peripheral neuropathy of Grade 2 or greater;
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel. Subjects with ulcerative colitis are also excluded;
* History of other malignancy. However, subjects who have been disease-free for 5 years, or subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma, are eligible;
* Concurrent disease or condition that would make the subject inappropriate for study participation, or any serious medical disorder that would interfere with the subject's safety;
* Uncontrolled infection;
* Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent;
* Known history of uncontrolled or symptomatic angina, arrhythmias, or congestive heart failure;
* Known history or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis;
* Concurrent treatment with prohibited medications, including herbal remedies and Chinese traditional medicines;
* Concurrent treatment with an investigational agent or participation in another clinical trial involving investigational agents;
* Used an investigational drug within 30 days or 5 half-lives, whichever is longer, preceding the first dose of investigational treatment;
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to paclitaxel or lapatinib or their excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 444 (Actual)
Dates: Start 2006-01-02 (Actual); Primary Completion 2010-06-18 (Actual); Study Completion 2021-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (38):
- Brazil (7):
  - Novartis Investigative Site, Salvador, Estado de Bahia
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Natal, Rio Grande do Norte
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Jaú, São Paulo
  - Novartis Investigative Site, Santo André, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- China (15):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Dalian, Liaoning
  - Novartis Investigative Site, Xi'an, Shaanxi
  - Novartis Investigative Site, Jinan, Shandong
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Chengdu
  - Novartis Investigative Site, Chongqing
  - Novartis Investigative Site, Dalian
  - Novartis Investigative Site, Fuzhou
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Shenyang
  - Novartis Investigative Site, Tianjin
- Hong Kong (3):
  - Novartis Investigative Site, Kowloon
  - Novartis Investigative Site, Pokfulam
  - Novartis Investigative Site, Tuenmen
- Novartis Investigative Site, Lahore, Pakistan
- Novartis Investigative Site, Lima, Peru
- Russia (5):
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Rostov-on-Don
  - Novartis Investigative Site, Samara
  - Novartis Investigative Site, Voronezh
- Thailand (2):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
- Ukraine (4):
  - Novartis Investigative Site, Cherkasy
  - Novartis Investigative Site, Chernihiv
  - Novartis Investigative Site, Dnipropetrovsk
  - Novartis Investigative Site, Zaporizhzhia

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Xu B, Guan Z, Shen Z, Tong Z, Jiang Z, Yang J, DeSilvio M, Russo M, Leigh M, Ellis C. Association of phosphatase and tensin homolog low and phosphatidylinositol 3-kinase catalytic subunit alpha gene mutations on outcome in human epidermal growth factor receptor 2-positive metastatic breast cancer patients treated with first-line lapatinib plus paclitaxel or paclitaxel alone. Breast Cancer Res. 2014 Jul 24;16(4):405. doi: 10.1186/s13058-014-0405-y. PMID 25056500
- [Derived] Guan Z, Xu B, DeSilvio ML, Shen Z, Arpornwirat W, Tong Z, Lorvidhaya V, Jiang Z, Yang J, Makhson A, Leung WL, Russo MW, Newstat B, Wang L, Chen G, Oliva C, Gomez H. Randomized trial of lapatinib versus placebo added to paclitaxel in the treatment of human epidermal growth factor receptor 2-overexpressing metastatic breast cancer. J Clin Oncol. 2013 Jun 1;31(16):1947-53. doi: 10.1200/JCO.2011.40.5241. Epub 2013 Mar 18. PMID 23509322
- See also: Related Info — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17997

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 43 centers in eight participating countries: Brazil (7), China (20), Hong Kong (3), Pakistan (3), Peru (1), Russian Federation (6), Thailand (2) and Ukraine (1).
Groups:
- Lapatinib 1500 mg + Paclitaxel: Lapatinib 1500 milligrams (mg) administered once daily plus paclitaxel 80 mg/meters squared (m^2) administered intravenously (IV) weekly for 3 weeks every 4 weeks
- Placebo + Paclitaxel: Matching placebo administered once daily plus paclitaxel 80 mg/m^2 administered IV weekly for 3 weeks every 4 weeks
- Open Label - Monotherapy: Open Label - Monotherapy (Lapatinib)
- Open Label - Combination Therapy: Open Label - Combination Therapy (Lapatinib and Paclitaxel)
Period: Randomized Phase
Arm/Group | Lapatinib 1500 mg + Paclitaxel | Placebo + Paclitaxel | Open Label - Monotherapy | Open Label - Combination Therapy
Started (All randomized subjects were included in the Intent-to-Treat (ITT) Population) | 222 | 222 | 0 | 0
Safety Population (All randomized subjects who received at least one dose of study medication) | 222 | 221 | 0 | 0
Completed | 133 | 149 | 0 | 0
Not Completed | 89 | 73 | 0 | 0
Not completed — Adverse Event | 0 | 2 | 0 | 0
Not completed — Lost to Follow-up | 34 | 27 | 0 | 0
Not completed — Withdrawal by Subject | 8 | 7 | 0 | 0
Not completed — Study closed/terminated | 1 | 1 | 0 | 0
Not completed — Disease progression | 36 | 27 | 0 | 0
Not completed — Physician Decision | 1 | 1 | 0 | 0
Not completed — Other reasons as defined per protocol | 4 | 3 | 0 | 0
Not completed — Reason for withdrawal unspecified | 4 | 5 | 0 | 0
Not completed — Treatment ongoing | 1 | 0 | 0 | 0
Period: Open Label Phase
Arm/Group | Lapatinib 1500 mg + Paclitaxel | Placebo + Paclitaxel | Open Label - Monotherapy | Open Label - Combination Therapy
Started | 0 | 0 | 149 | 4
Completed | 0 | 0 | 104 | 0
Not Completed | 0 | 0 | 45 | 4
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 16 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 2
Not completed — Disease progression | 0 | 0 | 18 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Relocation of patient | 0 | 0 | 1 | 0
Not completed — Reason for withdrawal unspecified | 0 | 0 | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lapatinib 1500 mg + Paclitaxel | Placebo + Paclitaxel | Total
Number analyzed (Participants) | 222 | 222 | 444
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.1 (10.74) | 49.3 (9.75) | 49.2 (10.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 222 | 217 | 439
  Male | 0 | 5 | 5
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 9 | 13 | 22
  Asian | 192 | 192 | 384
  Hispanic | 21 | 16 | 37
  Other | 0 | 1 | 1
Number of participants with any visceral metastatic disease and with only non-visceral disease [Count of Participants; unit: Participants] — Metastasis is defined as the spread of a tumor or cancerous cells from the primary site to one or more sites elsewhere in the body. Visceral metastasis is defined as the spread of cancer to viscera, the internal organs of the body, specifically those within the chest (as the heart or lungs) or abdomen (as the liver, pancreas, or intestines). Non-visceral organs are defined as any organ not considered visceral.
  Participants
    Visceral | 187 | 186 | 373
    Non-visceral | 35 | 36 | 71
Number of Participants with the Indicated Hormone Receptor Status [Count of Participants; unit: Participants] — Cancer cells have hormone receptor expression of Estrogen Receptor (ER) and/or Progesterone Receptor (PR) and are thus considered to be ER+ and/or PgR+ cells, respectively.
  Participants
    ER+ and/or PgR+ or Unknown | 111 | 113 | 224
    ER- and PgR- | 111 | 109 | 220
Number of Participants with the Indicated Stage of Disease at Initial Diagnosis [Count of Participants; unit: Participants] — The stage of cancer is a description of the extent to which the cancer has spread. Stage I cancer is localized; Stage II cancer has not started to spread into the surrounding tissue, but the tumor is larger than in Stage I; Stage III cancer is locally advanced and/or involves local lymph nodes; Stage IV cancer has spread to other organs.
  Participants
    Stage I to II | 107 | 119 | 226
    Stage III | 75 | 68 | 143
    Stage IV | 30 | 24 | 54
    Unknown | 10 | 11 | 21
Number of Participants with the Indicated Eastern Cooperative Oncology Group Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status classifies participants according to their functional impairment, and scores indicate: 0, fully active; 1, ambulatory, restricted strenuous activity; 2, ambulatory, no work activity; 3, partially confined to bed; 4, totally confined in bed; 5, death. Participants were required to have a baseline ECOG performance status of 0 or 1 for study participation.
  Participants
    0, Fully Active | 103 | 113 | 216
    1, Ambulatory, Restricted Strenuous Activity | 119 | 109 | 228
Number of Participants with the Indicated Number of Metastatic Sites [Count of Participants; unit: Participants] — Tumor cells move from the primary site to other sites in the body, where they continue to multiply and eventually form another clinically detectable tumor; thus, the site becomes metastatic. The table indicates number of metastatic sites.
  Participants
    Greater than or equal to 3 | 131 | 115 | 246
    Less than 3 | 91 | 107 | 198
Mean Time of Disease-Free Interval [Mean (Standard Deviation); unit: months] — The disease-free interval was defined as the time from initial diagnosis to metastases
  months | 27.51 (27.481) | 29.04 (34.522) | 28.27 (31.174)

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) at 53 Months
Description: Overall Survival (OS) was defined as the interval of time (in months) between the date of randomization and the date of death due to any cause.
Time Frame: From date of randomization until date of death from any cause, assessed up to 53 months (Primary OS analysis cut-off date = 18-Jun-2010)
Population: Intent-to-Treat (ITT) Population. The ITT population was comprised of all randomized subjects and was based on the treatment to which the subject was randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lapatinib 1500 mg + Paclitaxel | Placebo + Paclitaxel
Number analyzed (Participants) | 222 | 222
months | 27.8 [23.2 to 32.2] | 20.5 [17.9 to 24.3]
Statistical Analysis 1: Comparison: Lapatinib 1500 mg + Paclitaxel vs Placebo + Paclitaxel; Primary OS analysis cut-off date = 18-Jun-2010; Test type: Superiority or Other; p = 0.0062, Log Rank — Stratified Log-Rank (one-sided); Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.58 to 0.94] — The treatment hazard ratio based on the proportional hazard model stratifying for metastatic disease sites and hormonal status. A hazard ratio <1 indicates a lower risk with Lapatinib 1500mg + Paclitaxel compared with Placebo + Paclitaxel

2. Secondary Outcome: Overall Survival (OS) at 190 Months
Description: as for outcome 1
Time Frame: From date of randomization until date of death from any cause, assessed up to 190 months (Final OS analysis cut-off date = 23-Nov-2021)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lapatinib 1500 mg + Paclitaxel | Placebo + Paclitaxel
Number analyzed (Participants) | 222 | 222
months | 27.6 [23.7 to 31.5] | 20.3 [17.9 to 24.3]
Statistical Analysis 1: Comparison: Lapatinib 1500 mg + Paclitaxel vs Placebo + Paclitaxel; Final OS analysis cut-0ff date = 23-Nov-2021; Test type: Other; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.64 to 0.98] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Progression-free Survival (PFS) by Investigator Assessment
Description: Progression-free survival (PFS) during the randomized phase was defined as the interval of time (in months) between the date of randomization and the earlier of date of disease progression (radiological or clinical assessment of symptomatic progression), or date of death due to any cause.
Time Frame: From date of randomization until date of progression or date of death from any cause, whichever comes first, assessed up to 190 months (Final analysis cut-off date = 23-Nov-2021)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lapatinib 1500 mg + Paclitaxel | Placebo + Paclitaxel
Number analyzed (Participants) | 222 | 222
months | 9.7 [9.2 to 11.1] | 6.5 [5.5 to 7.3]
Statistical Analysis 1: Comparison: Lapatinib 1500 mg + Paclitaxel vs Placebo + Paclitaxel; Test type: Superiority or Other; Hazard Ratio (HR) = 0.54, 95% CI 2-sided [0.44 to 0.66] — The Pike estimator of the treatment hazard ratio based on the log rank test stratifying for metastatic disease sites and hormonal status. A hazard ratio <1 indicates a lower risk with Lapatinib 1500mg + Paclitaxel compared with Placebo + Paclitaxel

4. Secondary Outcome: Overall Response Rate (ORR) by Investigator Assessment
Description: Overall response rate (ORR) during the randomized phase was evaluated per Response Evaluation Criteria in Solid Tumors (RECIST v1.1) and defined as the percentage of subjects achieving either a Complete Response (CR) or a Partial Response (PR). Participants with unknown or missing responses were treated as non-responders.
Time Frame: From date of randomization until date of radiographic progression or date of death from any cause, whichever comes first, assessed up to 190 months (Final analysis cut-off date = 23-Nov-2021)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lapatinib 1500 mg + Paclitaxel | Placebo + Paclitaxel
Number analyzed (Participants) | 222 | 222
Percentage of Participants | 69 [62.9 to 75.4] | 50 [42.8 to 56.3]
Statistical Analysis 1: Comparison: Lapatinib 1500 mg + Paclitaxel vs Placebo + Paclitaxel; Test type: Superiority or Other; Odds Ratio (OR) = 2.30, 95% CI 2-sided [1.54 to 3.47]

5. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: Clinical benefit rate (CBR) was defined as the percentage of subjects with evidence of CR or PR or stable disease (neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of >=1 new lesions], taking as reference the smallest sum LD since treatment start) of >=24 weeks, based on confirmed responses from the investigator assessment of best overall response during the randomized phase.
Time Frame: From date of randomization until date of progression or date of death from any cause, whichever comes first, assessed up to 53 months (Primary analysis cut-off date = 18-Jun-2010)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lapatinib 1500 mg + Paclitaxel | Placebo + Paclitaxel
Number analyzed (Participants) | 222 | 222
Percentage of Participants | 75 [68.5 to 80.3] | 56 [49.1 to 62.5]
Statistical Analysis 1: Comparison: Lapatinib 1500 mg + Paclitaxel vs Placebo + Paclitaxel; Test type: Superiority or Other; Odds Ratio (OR) = 2.34, 95% CI 2-sided [1.54 to 3.58]

6. Secondary Outcome: Duration of Response (DOR)
Description: For subjects who show CR or PR, duration of response (DOR) was defined to be the time from first documented evidence of PR or CR until the first documented sign of disease progression (radiological or clinical assessment of symptomatic progression) or death due to any cause, if sooner during the randomized phase.
Time Frame: From date of confirmed CR or PR until date of progression or date of death from any cause, whichever comes first, assessed up to 190 months (Final analysis cut-off date = 23-Nov-2021)
Population: Subset of participants in the Intent-to-Treat (ITT) Population with a confirmed CR or PR
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lapatinib 1500 mg + Paclitaxel | Placebo + Paclitaxel
Number analyzed (Participants) | 154 | 110
months | 9.3 [7.7 to 10.7] | 5.8 [5.6 to 7.4]

7. Secondary Outcome: Number of Participants With a CR or PR at Weeks 8, 12, 16, 24, 32, 40, 48, 56, 64, and 72
Description: The original outcome measure to be analyzed was Time to response (TTR) during the randomized phase defined as the time from randomization until first documented evidence of PR or CR (whichever status was recorded first); however, data were presented as the number of participants with a response at each nominal visit. Responses were based on the investigator's assessment, and only participants with a confirmed CR or PR were included in this analysis.
Time Frame: Weeks 8, 12, 16, 24, 32, 40, 48, 56, 64, and 72
Population: Participants in the Intent-to-Treat (ITT) Population with a confirmed CR or PR
Measure: Number; unit: Participants
Arm/Group | Lapatinib 1500 mg + Paclitaxel | Placebo + Paclitaxel
Number analyzed (Participants) | 154 | 110
Participants
  Week 8 | 94 | 61
  Week 12 | 40 | 28
  Week 16 | 6 | 11
  Week 24 | 7 | 8
  Week 32 | 3 | 2
  Week 40 | 0 | 0
  Week 48 | 1 | 0
  Week 56 | 1 | 0
  Week 64 | 1 | 0
  Week 72 | 1 | 0

8. Secondary Outcome: Number of Tumors Evaluable for PIK3CA Mutations
Description: Phosphatidylinositol 3-kinase (PI3K) pathway deregulation (that is PIK3CA mutations and/or phosphatase and tensin homolog (PTEN) loss) was studied to evaluate the predictive and prognostic value of PIK3CA mutations and/or PTEN low in HER2-positive patients receiving first-line treatment with paclitaxel alone or in combination with lapatinib. A PIK3CA mutation test kit was used to assess mutation status on genomic deoxyribonucleic acid (DNA) isolated from tumor tissue.
Time Frame: Baseline
Population: Participants in the Intent-to-Treat (ITT) Population with tumors evaluable for PIK3CA mutations
Measure: Count of Participants; unit: Participants
Arm/Group | Lapatinib 1500 mg + Paclitaxel | Placebo + Paclitaxel
Number analyzed (Participants) | 104 | 106
Participants
  PIK3CA mutation | 29 | 36
  PIK3CA wild-type | 58 | 48
  PIK3CA indeterminate | 17 | 22

9. Secondary Outcome: Number of Participants With Tumors Evaluable for PTEN
Description: Phosphatidylinositol 3-kinase (PI3K) pathway deregulation (that is PIK3CA mutations and/or phosphatase and tensin homolog (PTEN) loss) was studied to evaluate the predictive and prognostic value of PIK3CA mutations and/or PTEN low in HER2-positive patients receiving first-line treatment with paclitaxel alone or in combination with lapatinib. Immunohistochemistry (IHC) staining in an analytically validated assay was used in the assessment of PTEN protein expression on tumor tissue. Staining intensity was allocated a score of 0, 1+, 2+ or 3+. Tumors scored IHC 0 were considered as exhibiting an absence of PTEN expression whereas those scored ICH 1+, 2+ or 3+ were considered as exhibiting any PTEN expression, being 3+ the highest expression.
Time Frame: Baseline
Population: Participants in the Intent-to-Treat (ITT) Population with tumors evaluable for PTEN
Measure: Count of Participants; unit: Participants
Arm/Group | Lapatinib 1500 mg + Paclitaxel | Placebo + Paclitaxel
Number analyzed (Participants) | 180 | 175
Participants
  PTEN IHC 0 | 28 | 21
  PTEN IHC 1+ | 76 | 80
  PTEN IHC 2+/3+ | 76 | 74

10. Secondary Outcome: Predictive Effect of PIK3CA Mutations Status on Overall Response Rate (ORR)
Description: ORR was evaluated per RECIST v1.1 and defined as the percentage of subjects achieving either CR or PR. Phosphatidylinositol 3-kinase (PI3K) pathway deregulation (that is PIK3CA mutations and/or phosphatase and tensin homolog (PTEN) loss) was studied to evaluate the predictive and prognostic value of PIK3CA mutations and/or PTEN low in HER2-positive patients receiving first-line treatment with paclitaxel alone or in combination with lapatinib. A PIK3CA mutation test kit was used to assess mutation status on genomic deoxyribonucleic acid (DNA) isolated from tumor tissue.
Time Frame: From date of randomization until date of radiographic progression or date of death from any cause, whichever comes first, assessed up to 53 months (Primary OS analysis cut-off date = 18-Jun-2010)
Population: Participants in the Intent-to-Treat (ITT) Population with tumors evaluable for PIK3CA mutations (PIK3CA mutation and PIK3CA wild type)
Measure: Number; unit: percentage of participants
Arm/Group | Lapatinib 1500 mg + Paclitaxel | Placebo + Paclitaxel
Number analyzed (Participants) | 87 | 84
percentage of participants
  PIK3CA mutation: number analyzed (Participants) | 29 | 36
  PIK3CA mutation | 62 | 50
  PIK3CA wild-type: number analyzed (Participants) | 58 | 48
  PIK3CA wild-type | 80 | 59
Statistical Analysis 1: Comparison: Lapatinib 1500 mg + Paclitaxel vs Placebo + Paclitaxel; Participants with PIK3CA wild-type; Test type: Other; Odds Ratio (OR) = 2.78, 95% CI 2-sided [1.07 to 7.57]

11. Secondary Outcome: Predictive Effect of PTEN Low on Overall Response Rate (ORR)
Description: ORR was evaluated per RECIST v1.1 and defined as the percentage of subjects achieving either CR or PR. Phosphatidylinositol 3-kinase (PI3K) pathway deregulation (that is PIK3CA mutations and/or phosphatase and tensin homolog (PTEN) loss) was studied to evaluate the predictive and prognostic value of PIK3CA mutations and/or PTEN low in HER2-positive patients receiving first-line treatment with paclitaxel alone or in combination with lapatinib. Immunohistochemistry (IHC) staining in an analytically validated assay was used in the assessment of PTEN protein expression on tumor tissue. Staining intensity was allocated a score of 0, 1+, 2+ or 3+. Tumors scored IHC 0 were considered as exhibiting an absence of PTEN expression whereas those scored ICH 1+, 2+ or 3+ were considered as exhibiting any PTEN expression, being 3+ the highest expression. Tumors scored IHC 0/1+ were considered PTEN low.
Time Frame: as for outcome 10
Population: Participants in the Intent-to-Treat (ITT) Population with PTEN low and without PTEN low
Measure: Number; unit: percentage of participants
Arm/Group | Lapatinib 1500 mg + Paclitaxel | Placebo + Paclitaxel
Number analyzed (Participants) | 180 | 175
percentage of participants
  PTEN low: number analyzed (Participants) | 104 | 101
  PTEN low | 73 | 53
  Without PTEN low: number analyzed (Participants) | 76 | 74
  Without PTEN low | 76 | 58
Statistical Analysis 1: Comparison: Lapatinib 1500 mg + Paclitaxel vs Placebo + Paclitaxel; Participants with PTEN low; Test type: Other; Odds Ratio (OR) = 2.42, 95% CI 2-sided [1.28 to 4.63]
Statistical Analysis 2: Comparison: Lapatinib 1500 mg + Paclitaxel vs Placebo + Paclitaxel; Participants without PTEN low; Test type: Other; Odds Ratio (OR) = 2.21, 95% CI 2-sided [1.04 to 4.82]

12. Secondary Outcome: Predictive Effect of PIK3CA Mutations Status on Clinical Benefit Rate (CBR)
Description: CBR was evaluated per RECIST v1.1 and defined as the percentage of subjects achieving CR or PR or stable disease. Phosphatidylinositol 3-kinase (PI3K) pathway deregulation (that is PIK3CA mutations and/or phosphatase and tensin homolog (PTEN) loss) was studied to evaluate the predictive and prognostic value of PIK3CA mutations and/or PTEN low in HER2-positive patients receiving first-line treatment with paclitaxel alone or in combination with lapatinib. A PIK3CA mutation test kit was used to assess mutation status on genomic deoxyribonucleic acid (DNA) isolated from tumor tissue.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Lapatinib 1500 mg + Paclitaxel | Placebo + Paclitaxel
Number analyzed (Participants) | 87 | 84
percentage of participants
  PIK3CA mutation: number analyzed (Participants) | 29 | 36
  PIK3CA mutation | 69 | 56
  PIK3CA wild-type: number analyzed (Participants) | 58 | 48
  PIK3CA wild-type | 84 | 65

13. Secondary Outcome: Predictive Effect of PTEN Low on Clinical Benefit Rate (CBR)
Description: CBR was evaluated per RECIST v1.1 and defined as the percentage of subjects achieving CR or PR or stable disease. Phosphatidylinositol 3-kinase (PI3K) pathway deregulation (that is PIK3CA mutations and/or phosphatase and tensin homolog (PTEN) loss) was studied to evaluate the predictive and prognostic value of PIK3CA mutations and/or PTEN low in HER2-positive patients receiving first-line treatment with paclitaxel alone or in combination with lapatinib. Immunohistochemistry (IHC) staining in an analytically validated assay was used in the assessment of PTEN protein expression on tumor tissue. Staining intensity was allocated a score of 0, 1+, 2+ or 3+. Tumors scored IHC 0 were considered as exhibiting an absence of PTEN expression whereas those scored ICH 1+, 2+ or 3+ were considered as exhibiting any PTEN expression, being 3+ the highest expression. Tumors scored IHC 0/1+ were considered PTEN low.
Time Frame: as for outcome 10
Population: Participants in the Intent-to-Treat (ITT) Population with PTEN low and without PTEN low
Measure: Number; unit: percentage of participants
Arm/Group | Lapatinib 1500 mg + Paclitaxel | Placebo + Paclitaxel
Number analyzed (Participants) | 180 | 175
percentage of participants
  PTEN low: number analyzed (Participants) | 104 | 101
  PTEN low | 82 | 59
  Without PTEN low: number analyzed (Participants) | 76 | 74
  Without PTEN low | 80 | 61
Statistical Analysis 1: Comparison: Lapatinib 1500 mg + Paclitaxel vs Placebo + Paclitaxel; Participants with PTEN low; Test type: Other; Odds Ratio (OR) = 3.15, 95% CI 2-sided [1.58 to 6.49]
Statistical Analysis 2: Comparison: Lapatinib 1500 mg + Paclitaxel vs Placebo + Paclitaxel; Participants without PTEN low; Test type: Other; Odds Ratio (OR) = 2.49, 95% CI 2-sided [1.13 to 5.66]

ADVERSE EVENTS:
Time Frame: From study treatment start date till 30 days safety follow-up, assessed up to 190 months (Final OS analysis cut-off date = 23-Nov-2021)
Description: Any sign or symptom that occurs during the treatment period plus 30 days post-treatment. The safety analysis were done on the safety population, which included all randomized subjects who received at least one dose of study medication.
Arm/Group | Lapatinib 1500 mg + Paclitaxel | Placebo + Paclitaxel | Open Label - Monotherapy | Open Label - Combination Therapy
All-Cause Mortality (participants affected / at risk) | 10/222 | 15/221 | 2/149 | 0/4
Serious Adverse Events (participants affected / at risk) | 67/222 | 30/221 | 8/149 | 0/4
Other Adverse Events (participants affected / at risk) | 219/222 | 206/221 | 86/149 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib 1500 mg + Paclitaxel (N=222) | Placebo + Paclitaxel (N=221) | Open Label - Monotherapy (N=149) | Open Label - Combination Therapy (N=4)
Febrile neutropenia (Blood and lymphatic system disorders) | 6 | 1 | 0 | 0
Granulocytopenia (Blood and lymphatic system disorders) | 4 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 7 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 36 | 10 | 0 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 1 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 3 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 10 | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0
Lithiasis (General disorders) | 1 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 3 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 1 | 0
Hepatobiliary disease (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Ejection fraction decreased (Investigations) | 13 | 3 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Intracranial pressure increased (Nervous system disorders) | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib 1500 mg + Paclitaxel (N=222) | Placebo + Paclitaxel (N=221) | Open Label - Monotherapy (N=149) | Open Label - Combination Therapy (N=4)
Anaemia (Blood and lymphatic system disorders) | 50 | 22 | 3 | 0
Granulocytopenia (Blood and lymphatic system disorders) | 17 | 15 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 113 | 74 | 6 | 0
Neutropenia (Blood and lymphatic system disorders) | 168 | 103 | 5 | 0
Abdominal distension (Gastrointestinal disorders) | 12 | 3 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 17 | 10 | 5 | 0
Abdominal pain upper (Gastrointestinal disorders) | 13 | 3 | 1 | 0
Constipation (Gastrointestinal disorders) | 8 | 18 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 172 | 64 | 42 | 0
Mouth ulceration (Gastrointestinal disorders) | 16 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 66 | 44 | 4 | 0
Vomiting (Gastrointestinal disorders) | 48 | 26 | 4 | 0
Asthenia (General disorders) | 15 | 7 | 1 | 0
Fatigue (General disorders) | 47 | 35 | 2 | 0
Mucosal erosion (General disorders) | 0 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 18 | 3 | 2 | 0
Oedema peripheral (General disorders) | 9 | 12 | 1 | 0
Pyrexia (General disorders) | 30 | 34 | 5 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 17 | 9 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 12 | 2 | 1 | 0
Paronychia (Infections and infestations) | 17 | 1 | 6 | 0
Upper respiratory tract infection (Infections and infestations) | 20 | 12 | 1 | 0
Alanine aminotransferase increased (Investigations) | 25 | 17 | 3 | 0
Aspartate aminotransferase increased (Investigations) | 20 | 16 | 4 | 0
Blood bilirubin increased (Investigations) | 7 | 5 | 2 | 1
Haemoglobin decreased (Investigations) | 23 | 4 | 0 | 0
Neutrophil count decreased (Investigations) | 3 | 1 | 0 | 1
Red blood cell count decreased (Investigations) | 6 | 1 | 0 | 1
White blood cell count decreased (Investigations) | 11 | 11 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 70 | 41 | 3 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 6 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 26 | 20 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 30 | 26 | 1 | 0
Dizziness (Nervous system disorders) | 19 | 11 | 0 | 0
Headache (Nervous system disorders) | 20 | 20 | 4 | 0
Hypoaesthesia (Nervous system disorders) | 18 | 25 | 3 | 0
Neuropathy peripheral (Nervous system disorders) | 31 | 30 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 12 | 13 | 0 | 0
Insomnia (Psychiatric disorders) | 13 | 18 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 22 | 22 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 | 12 | 2 | 0
Acne (Skin and subcutaneous tissue disorders) | 16 | 5 | 4 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 104 | 119 | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 16 | 3 | 8 | 2
Nail disorder (Skin and subcutaneous tissue disorders) | 26 | 3 | 8 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 23 | 9 | 10 | 0
Rash (Skin and subcutaneous tissue disorders) | 109 | 47 | 52 | 0

LIMITATIONS AND CAVEATS:
The data collected for China patients after 01JUL2019 were excluded from analysis due to local regulations in China.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.